CLINICAL TRIAL: NCT04259606
Title: Effect of Cassia Cinnamon on Arterial Stiffness Parameters in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Sara Pascoe Gonzalez, Principal investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCRA
Record Dates: First submitted 2019-10-23; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Arterial Stiffness
Keywords: Cassia cinnamon; Endothelial function; Pulse wave velocity; Brachial - ankle index

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, double blind, with control group. The study consists in two groups assigned to take either cassia cinnamon or placebo. Both groups will be taken Metformin as first line therapy for type 2 diabetes mellitus
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cassia Cinnamon (Active Comparator): Cassia cinnamon, capsule of 1 gram each, taken every 8 hours before meals for 90 days.
  Interventions: Dietary Supplement: Cassia Cinnamon
- Calcined Magnesia (Placebo Comparator): Placebo consists in calcined magnesia, capsule of 1 gram each, taken every 8 hours before meals for 90 days.
  Interventions: Other: Calcined magnesia

INTERVENTIONS:
Dietary Supplement: Cassia Cinnamon — Reddish - brown to light brown, typical sweet and aromatic free flowing powder.
  Arms: Cassia Cinnamon
Other: Calcined magnesia — White, odor, color and flavorless thin powder.
  Arms: Calcined Magnesia

SUMMARY:
Type 2 diabetes mellitus is considered a serious public health problem that has been raising worldwide. In Mexico, it is an important cause of morbi - mortality and it´s characterized by hyperglycemia that promotes an increase of cardiovascular risk through the impairment of arterial stiffness and endothelial function, which, in a chronic manner promotes the development of micro and macrovascular complications.

Many nutraceuticals have been currently implemented aimed to improve glycemic control, and reduce cardiovascular risk and it´s complications, which results in a better quality of life in patients with type 2 diabetes mellitus.

Cassia cinnamon pulverized bark has demonstrated to have vasodilator effect independent of endothelial mechanisms, probably regulating calcium influx or release into or within the cell, the later demonstrated in mice.

DETAILED DESCRIPTION:
A randomized, placebo control group, double blind clinical trial. 30 patients (male or female) from 40 to 65 years old with type 2 diabetes mellitus, less than 1 year of diagnosis, taking Metformin 850 mg daily, referred to the Experimental and Clinical Therapeutic Institute will be included.

All patients should give written informed consent prior to be enrolled. The protocol was previously approved by the local ethics committee (Experimental and Clinical Therapeutic Institute) of University of Guadalajara, registration number: CEI/489/2019. Patients with other medical conditions, taking additional drugs or with more than 1 year of evolution will be excluded.

Procedure:

The entire study consists of a total of 5 visits, the first one (day - 7) is the screening visit where written informed consent, clinical history, anthropometric measurements and blood samples will be performed.

The second or initial visit (day 0) consists of review of laboratory results, hemodynamic studies (i.e brachial - ankle pulse wave velocity and index for arterial stiffness and flow mediated dilation on brachial artery for endothelial function with VP1000 and UNEX EF devices respectively), and after randomization, start of intervention (either cassia cinnamon or placebo).

The third and fourth visits (day 30 and 60) consist of evaluation of treatment adherence, side effects, blood tests, treatment renewal and general recommendations.

The fifth and last visit (day 90) is similar to day 0 plus evaluation of treatment adherence and side effects. This is the end of intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to the beginning of enrollment
* Men and women 40 to 65 years old
* Diagnosis of type 2 diabetes mellitus according to the American Diabetes Association criteria
* Fasting plasma glucose ≥ 126 mg/dl (7.0 mmol/L) at least 8 h of fasting
* Plasma glucose ≥ 200 mg/dl (11.1 mmol/L) 2 hours after oral glucose tolerance test
* HbA1c ≥ 6.5 % (48 mmol/mol)
* Plasma glucose ≥ 200 mg/dl (11.1 mmol/L) in a random glucose test with typical symptoms of hyperglucemia or hyperglycemic crisis.

Exclusion Criteria:

* HbA1c < 6.5 % or > 10 % or fasting glucose plasma > 250 mg/dl
* Total serum cholesterol ≥ 240 mg/dl
* Triglycerides ≥ 400 mg/dl
* History of allergy to any of the components used in the study
* Consumption of additional drugs with known effects on glucose and lipids metabolism and weight reduction
* History of cardiovascular disease, blood abnormalities and/or kidney, pancreatic or thyroid disease
* Childbearing and breastfeeding women
* History of smoking within 12 months prior to beginning of study
* History of drug abuse and alcoholism
* Pacemaker bearing or any other permanent bioelectronic device that could modify or interfere with electrical bioimpedance tests

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Brachial - ankle pulse wave velocity | 90 days
  Change in the pulse wave velocity
Flow mediated dilation | 90 days
  Change in the capacity of dilation of the brachial artery
Brachial - ankle index | 90 days
  Change in the systolic and diastolic pressures of the brachial and tibial arteries, the index is the result of dividing the last between the first

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | 4 visits: days 1, 30, 60 and 90.
  Millimeters of mercury. mmHg
Blood glucose | 4 visits: days 1, 30, 60 and 90.
  Milligrams over deciliters. mg/dL
Glycated hemoglobin | 4 visits: days 1, 30, 60 and 90.
  Percentage
Lipid profile | 4 visits: days 1, 30, 60 and 90.
  Total cholesterol, triglycerides, high density lipoprotein, very high density lipoprotein, low density lipoprotein. All of them expressed in milligrams over deciliters. mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Ofelia Hernández González, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2019 Abridged for Primary Care Providers. Clin Diabetes. 2019 Jan;37(1):11-34. doi: 10.2337/cd18-0105. No abstract available. PMID 30705493
- [Background] Rosas Y, Calles J. Documento de posición de la Asociación Latinoamericana de Diabetes (ALAD). Consenso de prediabetes. 2009;17:146-158
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Arauz A, Ruíz-Franco A. Enfermedad Vascular Cerebral. Rev Fac Medicina UNAM.2012;55:11-21
- [Background] Ritz E. Nephropathy in type 2 diabetes. J Intern Med. 1999 Feb;245(2):111-26. doi: 10.1046/j.1365-2796.1999.00411.x. PMID 10081514
- [Background] Javed S, Alam U, Malik RA. Treating Diabetic Neuropathy: Present Strategies and Emerging Solutions. Rev Diabet Stud. 2015 Spring-Summer;12(1-2):63-83. doi: 10.1900/RDS.2015.12.63. Epub 2015 Aug 10. PMID 26676662
- [Background] Pedraza L. Neuropatías diabéticas, formas clínicas y diagnóstico. Rev Med Clin.2009;20:681-686
- [Background] Julio R, Galleguillos I. Diabetes y enfermedad vascular periférica. Rev Med Clin. 2009;20:687-697
- [Background] Cervantes R, Presno J. Fisiopatología de la diabetes y los mecanismos de muerte de las células β pancreáticas. Rev. Endocrinol. Nutr.2013;21:98-106
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Background] DeFronzo RA, Abdul-Ghani M. Type 2 diabetes can be prevented with early pharmacological intervention. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S202-9. doi: 10.2337/dc11-s221. PMID 21525456
- [Background] de Oliveira Alvim R, Santos PCJL, Musso MM, de Sa Cunha R, Krieger JE, Mill JG, Pereira AC. Impact of diabetes mellitus on arterial stiffness in a representative sample of an urban Brazilian population. Diabetol Metab Syndr. 2013 Aug 21;5(1):45. doi: 10.1186/1758-5996-5-45. PMID 23965633
- [Background] Jia G, Aroor AR, DeMarco VG, Martinez-Lemus LA, Meininger GA, Sowers JR. Vascular stiffness in insulin resistance and obesity. Front Physiol. 2015 Aug 14;6:231. doi: 10.3389/fphys.2015.00231. eCollection 2015. PMID 26321962
- [Background] Yeboah K, Antwi DA, Gyan B. Arterial Stiffness in Nonhypertensive Type 2 Diabetes Patients in Ghana. Int J Endocrinol. 2016;2016:6107572. doi: 10.1155/2016/6107572. Epub 2016 Sep 28. PMID 27774104
- [Background] Li X, Deng YP, Yang M, Wu YW, Sun SX, Sun JZ. Low-Grade Inflammation and Increased Arterial Stiffness in Chinese Youth and Adolescents with Newly-Diagnosed Type 2 Diabetes Mellitus. J Clin Res Pediatr Endocrinol. 2015 Dec;7(4):268-73. doi: 10.4274/jcrpe.2187. PMID 26777037
- [Background] Morales S, Garcia-Salcedo JA, Munoz-Torres M. [Pentosidine: a new biomarker in diabetes mellitus complications]. Med Clin (Barc). 2011 Mar 19;136(7):298-302. doi: 10.1016/j.medcli.2009.12.001. Epub 2010 Mar 11. Spanish. PMID 20226481
- [Background] Cardoso CR, Salles GF. Aortic Stiffness as a Surrogate Endpoint to Micro- and Macrovascular Complications in Patients with Type 2 Diabetes. Int J Mol Sci. 2016 Dec 6;17(12):2044. doi: 10.3390/ijms17122044. PMID 27929441
- [Background] Weisbrod RM, Shiang T, Al Sayah L, Fry JL, Bajpai S, Reinhart-King CA, Lob HE, Santhanam L, Mitchell G, Cohen RA, Seta F. Arterial stiffening precedes systolic hypertension in diet-induced obesity. Hypertension. 2013 Dec;62(6):1105-10. doi: 10.1161/HYPERTENSIONAHA.113.01744. Epub 2013 Sep 23. PMID 24060894
- [Background] Townsend RR, Wilkinson IB, Schiffrin EL, Avolio AP, Chirinos JA, Cockcroft JR, Heffernan KS, Lakatta EG, McEniery CM, Mitchell GF, Najjar SS, Nichols WW, Urbina EM, Weber T; American Heart Association Council on Hypertension. Recommendations for Improving and Standardizing Vascular Research on Arterial Stiffness: A Scientific Statement From the American Heart Association. Hypertension. 2015 Sep;66(3):698-722. doi: 10.1161/HYP.0000000000000033. Epub 2015 Jul 9. No abstract available. PMID 26160955
- [Background] Suarez C, Ruilope LM. [New guidelines from the World Health Organization and the International Society of Hypertension for the management of hypertension: toward common guidelines]. Rev Esp Cardiol. 1999 Jun;52(6):381-2. doi: 10.1016/s0300-8932(99)74934-1. No abstract available. Spanish. PMID 10373770
- [Background] Medagama AB, Bandara R. The use of complementary and alternative medicines (CAMs) in the treatment of diabetes mellitus: is continued use safe and effective? Nutr J. 2014 Oct 21;13:102. doi: 10.1186/1475-2891-13-102. PMID 25331834
- [Background] Chang CT, Chang WL, Hsu JC, Shih Y, Chou ST. Chemical composition and tyrosinase inhibitory activity of Cinnamomum cassia essential oil. Bot Stud. 2013 Dec;54(1):10. doi: 10.1186/1999-3110-54-10. Epub 2013 Aug 21. PMID 28510850
- [Background] Rao PV, Gan SH. Cinnamon: a multifaceted medicinal plant. Evid Based Complement Alternat Med. 2014;2014:642942. doi: 10.1155/2014/642942. Epub 2014 Apr 10. PMID 24817901
- [Background] Vangalapati M, Satya S, Prakash S, Avanigadda S. A review on pharmacological activities and clinical effects of Cinnamon species. J Pharm Biol Chem Sci. 2012;3(1):653-663
- [Background] Akilen R, Tsiami A, Devendra D, Robinson N. Glycated haemoglobin and blood pressure-lowering effect of cinnamon in multi-ethnic Type 2 diabetic patients in the UK: a randomized, placebo-controlled, double-blind clinical trial. Diabet Med. 2010 Oct;27(10):1159-67. doi: 10.1111/j.1464-5491.2010.03079.x. PMID 20854384
- [Background] Xue YL, Shi HX, Murad F, Bian K. Vasodilatory effects of cinnamaldehyde and its mechanism of action in the rat aorta. Vasc Health Risk Manag. 2011;7:273-80. doi: 10.2147/VHRM.S15429. Epub 2011 Apr 28. PMID 21603596
- [Background] Kang YH, Yang IJ, Morgan KG, Shin HM. Cinnamyl alcohol attenuates vasoconstriction by activation of K(+) channels via NO-cGMP-protein kinase G pathway and inhibition of Rho-kinase. Exp Mol Med. 2012 Dec 31;44(12):749-55. doi: 10.3858/emm.2012.44.12.083. PMID 23178275
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804
- [Background] Ziegenfuss TN, Hofheins JE, Mendel RW, Landis J, Anderson RA. Effects of a water-soluble cinnamon extract on body composition and features of the metabolic syndrome in pre-diabetic men and women. J Int Soc Sports Nutr. 2006 Dec 28;3(2):45-53. doi: 10.1186/1550-2783-3-2-45. PMID 18500972
- [Background] Jeyaseelan L, Rao PS. Methods of determining sample sizes in clinical trials. Indian Pediatr. 1989 Feb;26(2):115-21. PMID 2753525
- [Background] Zócalo Y, Bia D. Presión aórtica central y parámetros clínicos derivados de la onda del pulso: evaluación no invasiva en la práctica clínica. Rev Urug Cardiol. 2014;29:215-230
- [Background] Gomez Marcos MA, Recio Rodriguez JI, Rodriguez Sanchez E, Patino Alonso MC, Gomez Sanchez L, Garcia ortiz L. [The increase in the speed of the pulse wave is not associated with elevated central blood pressure in hypertensive patients with kidney disease]. Nefrologia. 2010;30(5):578-83. doi: 10.3265/Nefrologia.pre2010.June.10383. Spanish. PMID 20613849
- [Background] Calabia Martínez, J. Medida de la Velocidad de Onda de Pulso mediante Ecografía Doppler: Concordancia con el Método Complior.2016
- [Background] Sáez J. Distensibilidad arterial: un parámetro más para valorar el riesgo cardiovascular. SEMERGEN. 2008;34(6):284-90
- [Background] Polo C, Del Castillo M. El índice cintura-cadera. Revisión. Madrid: Centro de Medicina Deportiva, Comunidad de Madrid
- [Background] Compendio de Leyes y Reglamentos. Agenda de Salud 2002. Tercera edición. México: Ediciones fiscals ISEF, 2002
- [Background] Rabkin SW, Chan SH, Sweeney C. Ankle-brachial index as an indicator of arterial stiffness in patients without peripheral artery disease. Angiology. 2012 Feb;63(2):150-4. doi: 10.1177/0003319711410307. Epub 2011 Jun 15. PMID 21676966
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Mozos I, Malainer C, Horbanczuk J, Gug C, Stoian D, Luca CT, Atanasov AG. Inflammatory Markers for Arterial Stiffness in Cardiovascular Diseases. Front Immunol. 2017 Aug 31;8:1058. doi: 10.3389/fimmu.2017.01058. eCollection 2017. PMID 28912780
- [Background] Hamilton SJ, Watts GF. Endothelial dysfunction in diabetes: pathogenesis, significance, and treatment. Rev Diabet Stud. 2013 Summer-Fall;10(2-3):133-56. doi: 10.1900/RDS.2013.10.133. Epub 2013 Aug 10. PMID 24380089
- [Background] Bia D, Zócalo Y. Rigidez arterial: evaluación no invasiva en la práctica clínica. Rev Urug Cardiol. 2014;29:39-59
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] Christen A, Miranda A, Caride S, Armentano R, Ramírez A, Sánchez R. Velocidad de la onda de pulso: relevancia de la edad en normotensión, hipertensión escencial e hipertensión limítrofe. Rev. Argent. Cardiol. 2015;83:112-118
- [Background] Sánchez-Martínez M, Cruz J, Graciani A, García E, Artalejo F, Banegas J. Velocidad de la onda de pulso y presión arterial central: valores normales y de referencia en personas mayores en España. Rev Esp Cardiol. 2018:1-3
- [Background] Zhu R, Liu H, Liu C, Wang L, Ma R, Chen B, Li L, Niu J, Fu M, Zhang D, Gao S. Cinnamaldehyde in diabetes: A review of pharmacology, pharmacokinetics and safety. Pharmacol Res. 2017 Aug;122:78-89. doi: 10.1016/j.phrs.2017.05.019. Epub 2017 May 27. PMID 28559210
- [Background] Hajimonfarednejad M, Ostovar M, Raee MJ, Hashempur MH, Mayer JG, Heydari M. Cinnamon: A systematic review of adverse events. Clin Nutr. 2019 Apr;38(2):594-602. doi: 10.1016/j.clnu.2018.03.013. Epub 2018 Apr 5. PMID 29661513
- [Background] Diabetes, O. M. S. Informe Mundial sobre la Diabetes. Ginebra. 2016
- [Background] Instituto Nacional de Estadística y Geografía. Principales causas de mortalidad por residencia habitual, grupos de edad y sexo del fallecido. 2016
- [Background] International Diabetes Federation. IDF Diabetes Atlas. 8ª edición. 2017
- [Background] Romero-Martinez M, Shamah-Levy T, Cuevas-Nasu L, Gomez-Humaran IM, Gaona-Pineda EB, Gomez-Acosta LM, Rivera-Dommarco JA, Hernandez-Avila M. [Methodological design of the National Health and Nutrition Survey 2016]. Salud Publica Mex. 2017 May-Jun;59(3):299-305. doi: 10.21149/8593. Spanish. PMID 28902317
- [Background] National Institute for Healt and Care Excellence. Type 2 diabetes: prevention in people at high risk. Pub. Health Guidel. 2012
- [Background] Prevención secundaria, diagnóstico, tratamiento y vigilancia de la enfermedad cerebral isquémica. México Secretaría de Salud. 2008
- [Background] Martinez-Murillo C, Aguilar-Arteaga ML, Velasco-Ortega E, Alonso-Gonzalez R, Castellanos-Sinco H, Romo-Jimenez A, Vargas-Ruiz A, Torres-Arreola L, Viniegra-Osorio A. [Clinical guideline for diagnosis and treatment of the thromboembolic venous disease]. Rev Med Inst Mex Seguro Soc. 2011 Jul-Aug;49(4):437-49. Spanish. PMID 21982196
- [Background] Millan-Gamez YK, Wacher-Rodarte NH, Bravo-Ortiz JC, Garrido-Gaspar NH, Mendoza-Topete R, Martinez-Ruiz AM, Miller-Arrevillaga G, Ramirez-Najera A. [Clinical practice guidelines. Diagnosis and treatment of diabetic retinopathy]. Rev Med Inst Mex Seguro Soc. 2011 Sep-Oct;49(5):551-62. Spanish. PMID 22185860
- [Background] Harrison´s Principles of Internal Medicine (2015). Kasper D, Hauser S, Jameson J. McGrawHill
- [Background] Herbs & natural supplements an evidence-based guide. 2010. Braun L, Cohen M. ELSEVIER
- [Derived] Delgadillo-Centeno JS, Grover-Paez F, Hernandez-Gonzalez SO, Ramos-Zavala MG, Cardona-Muller D, Lopez-Castro A, Pascoe-Gonzalez S. Cinnamomum cassia on Arterial Stiffness and Endothelial Dysfunction in Type 2 Diabetes Mellitus: Outcomes of a Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Med Food. 2023 Jun;26(6):428-434. doi: 10.1089/jmf.2022.0089. Epub 2023 Jun 1. PMID 37262194
- See also: Chemical properties of bark cinnamon derived Cinnamaldehyde — http://pubchem.ncbi.nlm.nih.gov